CLINICAL TRIAL: NCT07230301
Title: Intracavitary Infusion of Adebrelimab Combined With the Best Standard Treatment for the Treatment of Pancreatic Cancer With Pleural and Peritoneal Effusions: A Single-Center, Prospective, Clinical Trial
Brief Title: Adebrelimab Infusion Plus Standard Care for Pancreatic Cancer With Pleural or Peritoneal Effusions
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sizhen Wang (Other)
Responsible Party: Sponsor-Investigator, Sizhen Wang, Chief Physician / Professor, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZQH-KYLLFS-25-19
Record Dates: First submitted 2025-09-28; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer Metastatic
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: This is a single-center, single-arm, prospective Phase II interventional study. All enrolled patients receive intracavitary infusion of adebrelimab combined with investigator's choice of best supportive treatment. The model is designed to evaluate safety and efficacy without a control arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Adebrelimab 600 mg administered intrapleurally or intraperitoneally on Days 1 and 8 of each 3-week cycle (Q3W), combined with investigator's choice of best supportive care (chemotherapy or targeted agents). Administration continues even if effusion decreases or becomes non-drainable.
  Interventions: Drug: Adebrelimab (PD-L1 inhibitor)

INTERVENTIONS:
Drug: Adebrelimab (PD-L1 inhibitor) — Adebrelimab 600 mg administered by intrapleural or intraperitoneal infusion on Days 1 and 8 of each 3-week cycle (Q3W). Treatment is combined with investigator's choice of best supportive therapy, such as chemotherapy or targeted agents. Administration continues even if effusion decreases or becomes non-drainable.

SUMMARY:
1. Study:

   A Clinical Study of Intra-cavity Adebrelimab Combined with Best Supportive Care for Pancreatic Cancer Patients with Pleural or Peritoneal Effusion (Malignant Ascites)
2. Why is this study being done? This study is being done to find out if a new approach to treatment is safe and effective for controlling malignant fluid buildup (pleural or peritoneal effusion) in the abdomen or chest in patients with pancreatic cancer. The approach involves putting a drug called Adebrelimab directly into the fluid cavity, in combination with the best available supportive care chosen by your doctor.
3. What is Adebrelimab? Adebrelimab is a type of immunotherapy drug (a PD-L1 inhibitor) that helps the body's immune system fight cancer cells. It is already approved in China for treating some lung cancers. In this study, it is being given directly into the fluid buildup (intra-cavity) to see if it can work better there.
4. What will happen if I join the study?

   Screening: First, you will go through tests to see if you are eligible.

   Treatment: If eligible, the fluid will be drained. Then, Adebrelimab will be infused into the cavity on Day 1 and Day 8 of each 3-week cycle. You will also receive the best supportive care for your cancer.

   Monitoring: You will have regular clinic visits for check-ups, blood tests, and scans to see how you are responding to the treatment and to monitor for any side effects.
5. How long will I be in the study? Treatment will continue as long as it is controlling the disease, you are not experiencing unacceptable side effects, and you choose to remain in the study.
6. What are the potential benefits? You may experience a reduction in the cancer-related fluid buildup and better control of your cancer. However, benefit cannot be guaranteed. The information from this study may also help other patients in the future.
7. What are the potential risks and side effects? Possible side effects of Adebrelimab include nausea, fatigue, decreased appetite, vomiting, diarrhea, low blood cell counts, and abnormal liver tests. There may also be unknown risks. The best supportive care has its own risks, which your doctor will explain. You will be monitored closely for safety.
8. What are my other choices? You can choose not to participate. This will not affect your standard medical care. Your other options may include drainage of the fluid and other standard treatments aimed at managing your symptoms and cancer.
9. Is participation voluntary? Yes. Your participation is completely voluntary. You can decide to leave the study at any time, for any reason, without any penalty or loss of benefits to which you are entitled.

DETAILED DESCRIPTION:
Patients with pancreatic cancer and malignant pleural or peritoneal effusions first undergo screening, including imaging, laboratory tests, and confirmation of malignant effusion. After informed consent and baseline assessments, they receive intracavitary infusion of adebrelimab (600 mg on days 1 and 8 of each 3-week cycle), combined with the investigator's choice of best supportive treatment such as chemotherapy or targeted therapy. Even if effusion is markedly reduced or drainage becomes impossible, intracavitary administration is continued. Clinical monitoring involves regular vital signs, laboratory evaluations, and recording of adverse events according to NCI-CTCAE v5.0.

Efficacy is assessed by imaging every six weeks and ultrasound measurement of effusion volume, with treatment responses categorized as complete response, partial response, stable disease, or progression. The primary endpoint is overall survival, while secondary endpoints include objective response rate, progression-free survival, disease control rate, puncture-free survival, and effusion control rate. After the last dose, patients enter a 30-day safety follow-up, and then survival status is checked every 90 days until death or loss to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.

Histologically or cytologically confirmed pancreatic cancer.

Presence of malignant pleural or peritoneal effusion (≥4 cm) confirmed by pathology or cytology, requiring clinical intervention.

At least one measurable lesion according to RECIST v1.1.

ECOG performance status 0-3.

Estimated life expectancy ≥ 2 months.

Adequate organ function:

Hemoglobin ≥ 80 g/L

ANC ≥ 1.0 × 10⁹/L

Platelets ≥ 50 × 10⁹/L

TBIL < 3 × ULN

ALT/AST < 5 × ULN

Serum creatinine ≤ 1.25 × ULN or creatinine clearance > 45 mL/min

Chronic HBV infection must be controlled with antiviral therapy and HBV DNA < 10,000 IU/mL.

Women of childbearing potential must have a negative pregnancy test and agree to use effective contraception during the study and for at least 8 weeks after the last dose; men must agree to contraception or have undergone sterilization.

Voluntarily signed informed consent with good compliance for follow-up.

Exclusion Criteria:

* Asymptomatic effusion not requiring intervention.

Contraindication to paracentesis or drainage.

Contraindications to immunotherapy (e.g., chronic steroid use, prior immune-related pneumonitis, hepatitis, or colitis).

Active autoimmune disease requiring systemic therapy.

Active HCV, HIV, syphilis, or tuberculosis infection; uncontrolled severe infection within 4 weeks prior to first dose.

History of allogeneic organ transplantation or autologous stem cell transplantation.

Severe pulmonary disease (e.g., pulmonary fibrosis, interstitial lung disease, pneumoconiosis).

History of psychiatric illness or substance abuse affecting compliance.

Participation in another interventional clinical trial within 4 weeks.

Prior treatment with PD-1/PD-L1 antibodies via intrapleural or intraperitoneal route.

Uncontrolled CNS metastases or intracranial hypertension.

Active bleeding tendency, GI bleeding within 4 weeks, or ongoing anticoagulation/thrombolysis therapy.

Other active malignancies (except cured basal cell carcinoma, cervical carcinoma in situ, or superficial bladder cancer).

Pregnant or breastfeeding women.

Any other condition judged by the investigator to affect participation or evaluation of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From first dose until death, assessed up to 36 months
  Time from first dose until death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From first dose until disease progression or death, assessed up to 36 months
  Proportion of patients achieving complete response (CR) or partial response (PR) per RECIST v1.1.
Progression-Free Survival (PFS) | From first dose until disease progression or death, assessed up to 36 months
  Time from the date of first dose of study treatment until the first documented disease progression per RECIST v1.1 or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | From first dose until disease progression, death, or last tumor assessment, assessed up to 36 months
  Proportion of patients achieving CR, PR, or stable disease (SD).
Puncture-Free Survival | From last dose until re-drainage of effusion or death, assessed up to 36 months
  Time from last dose until the need for re-drainage of effusion or death.
Effusion Control Rate | From first dose, assessed every 3 weeks until disease progression or death, up to 36 months
  Proportion of patients with complete or partial control of malignant pleural/peritoneal effusion.
Safety and Tolerability | From baseline through 90 days after the last dose of study treatment
  Incidence and severity of adverse events graded according to NCI-CTCAE v5.0.